CLINICAL TRIAL: NCT01351428
Title: Non-invasive Hemodynamic Monitoring and Goal-Directed Therapy in Pregnant Women at High Risk of Developing Preeclampsia
Brief Title: Goal-Directed Therapy in Pregnant Women at High Risk of Developing Preeclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-03
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Pre-Eclampsia; Pregnancy; Hypertension
Keywords: Non invasive cardiac output monitor; NICOM; Hypertension; Pregnancy; Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia; Hypertension | interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NICOM group (Experimental): Vasodilator therapy begins when SVR increases by 20% or greater than baseline. Therapy is titrated according to hemodynamic profile and clinical signs and symptoms.
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Nifedipine — 30-60 mg, twice daily
  Other Names: Adalat XL

SUMMARY:
Preeclampsia is associated with significant maternal and fetal morbidity and mortality. Early identification and subsequent management of patients at risk of developing preeclampsia presents an ongoing challenge in prenatal care. Some at risk pregnancies may be identified from:

* serum screening abnormalities in the first or second trimester
* placental shape and texture at the 18-20 anatomical ultrasound
* uterine artery blood flow.

Early identification and effective treatment of patients would permit the safe completion of the pregnancy for the mother and infant. Recent advances in non-invasive cardiovascular monitoring have enabled the study of maternal hemodynamics in normal and at-risk pregnancies. This study hopes to identify the earliest significant changes in maternal hemodynamics which may allow targeted therapeutic interventions in patients at high risk of developing preeclampsia.

The hypothesis of this study is that systemic vascular resistance rises during the pre-clinical phase of preeclampsia and this can be captured using non invasive bioreactance technology. Treatment of the abnormally high vascular tone may decrease the severity and postpone the onset of clinical disease.

DETAILED DESCRIPTION:
Invasive hemodynamic techniques have long identified significant increases in heart rate (HR), blood volume, left ventricular end-diastolic volume (LVEDV), stroke volume (SV) and cardiac output (CO) during the first and second trimesters of pregnancy. In normal pregnancy, CO increases from as early as 5 weeks gestation, with a 30-40% increase by the end of the first trimester of pregnancy. Cardiac output continues to rise throughout the second trimester until it reaches a level approximately 50% greater than that of non-pregnant women. Cardiac output slightly decreases during the third trimester. Despite these changes, maternal blood pressure (BP) still falls due to a large reduction in systemic vascular resistance (SVR) from systemic vasodilatation and the formation of a low-resistance utero-placental circulation. Systemic vascular resistance falls during early gestation, reaching its nadir (35% decline) at 20 weeks gestation, and rises during late pregnancy.

Transthoracic bioreactance is a newer technique of non-invasive continuous cardiac output monitoring. It is based on an analysis of relative phase shifts of oscillating currents that occur when this current traverses the thoracic cavity, as opposed to the traditional bioimpedance-based system, which rely only on measured changes in signal amplitude. Unlike bioimpedance, bioreactance-based non-invasive CO measurement does not use the static impedance and does not depend on the distance between the electrodes for the calculations of SV and CO, which significantly reduces the uncertainty in the result. Moreover, its readings were shown to correlate well with results derived from pulmonary artery catheter derived measurement of cardiac output. In addition, it has also been shown that the non-invasive cardiac output measurement (NICOM®) system has acceptable accuracy, precision and responsiveness for CO monitoring in patients experiencing a wide range of circulatory situations and has recently been used in the obstetric population.

The purpose of this study is to use non-invasive cardiac output monitoring to capture the earliest inappropriate rise in SVR during the pre clinical phase of disease, in patients at high risk of developing preeclampsia, as predicted by the placenta profile. In case an increase in SVR is identified, the purpose of this study is to implement a goal-directed therapy in an attempt to decrease the severity, and postpone the onset of clinical disease.

The hypothesis of this study is that the increases in SVR detected during the pre-clinical phase of preeclampsia can be treated with a goal directed therapy without fetal compromise and that this intervention may improve maternal and fetal/neonatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Risk factors for preeclampsia/IUGR - medical or obstetric
* Abnormal uterine artery Doppler
* Two of the following:

Abnormal placental biochemistry Abnormal placental shape Abnormal placental texture

Exclusion Criteria:

* Multifetal pregnancy
* Fetal abnormality, including nuchal translucency more than 3mm at 12 weeks
* Preterm labor/pprom/bleeding/rescue cerclage (excluding elective 12 week prophylactic cerclage)
* Type 1 diabetes mellitus
* Heparin use
* Chronic hypertension on treatment before 20 weeks
* Documented chronic renal disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Systemic vascular resistance | 20-22, 24-26, 28, 30-32 and 36 weeks gestational age
  Systemic vascular resistance is measured at the above time points, and more frequently at the discretion of the attending obstetrician.

SECONDARY OUTCOMES:
Maximum change in maternal blood pressure | 20-22, 24-26, 28, 30-32 and 36 weeks gestational age
  Blood pressure is taken on the NICOM at the above time points, and more frequently at obstetric appointments in between.
Gestational age at delivery | 25-41 weeks gestational age
Fetal weight at delivery | 25-41 weeks gestational age
Gestational age at time of first hospitalization | 25-41 weeks gestational age
Gestational age at peak maternal blood pressure | 20-41 weeks
Gestational age at which steroids are administered | 25-41 weeks gestational age
Serum s-Flt and PlGF levels | 12-41 weeks gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Jose CA Carvalho, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada